CLINICAL TRIAL: NCT03076723
Title: Using Cerebrospinal Fluid Dynamics to Identify Shunt Responders in Idiopathic Normal Pressure Hydrocephalus and to Optimize Postoperative Clinical Improvement While Minimizing Overdrainage Related Complications - A Double Blind Randomized Study
Brief Title: Using Cerebrospinal Fluid Dynamics to Optimize Treatment of Idiopathic Normal Pressure Hydrocephalus
Acronym: PULSE-OPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Acceptable duration exceeded. Enrolment too slow due to covid pandemic and extensive protocol.
Sponsor: Umeå University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Uppsala University Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMU-2016-CSFD-PC
Record Dates: First submitted 2016-12-13; First posted 2017-03-10 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Hydrocephalus, Normal Pressure
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed opening pressure (Sham Comparator): The shunt opening pressure is changed to the same setting as at surgery.
  Interventions: Other: Simulated change in shunt opening pressure
- Individual shunt opening pressure (Experimental): The shunt opening pressure is adjusted (up one step, down one step or unchanged) according to an individual analysis of the pulsatility curve (as assessed after shunt surgery).
  Interventions: Other: Change in shunt opening pressure

INTERVENTIONS:
Other: Change in shunt opening pressure — An individually determined change in shunt opening pressure is compared to no change in opening pressure.
  Arms: Individual shunt opening pressure
Other: Simulated change in shunt opening pressure — The shunt opening pressure is reset to the same setting.
  Arms: Fixed opening pressure

SUMMARY:
The purpose of the study is to determine if the so called pulsatility curve, which describes the relationship between intracranial pressure (ICP) and ICP pulsatility, can be used to predict outcome of treatment, in the form of shunt surgery, in idiopathic normal pressure hydrocephalus (INPH) and to guide the adjustment of shunt opening pressure after the surgery. The main hypotheses of the study are:

1. The pulsatility curve may be the best auxiliary test to predict shunt surgery outcome in INPH patients. With a "fixed" shunt opening pressure, the preoperatively assessed potential pulse amplitude reduction (determined by analysis of the pulsatility curve) predicts postoperative improvement in gait velocity and cognitive functions.
2. A postoperative pulsatility curve can be used to further optimize ICP pulsatility by guiding opening pressure adjustment. Shunt adjustment based on the pulsatility curve three months postoperatively will increase improvement, but not complications, compared to a shunt with "fixed" opening pressure.

Based on these hypotheses, three specific aims for the study have been defined:

1. To determine if improvement three month after surgery is associated with postoperative reduction in pulse amplitude.
2. To determine if a pulsatility curve obtained preoperatively can predict improvement in gait velocity and cognitive functions in INPH patients three months after surgery.
3. To compare outcome six months after surgery and complications rates between INPH patients with a "fixed" opening pressure versus those where the shunt has been adjusted based on the pulsatility curve, three months after the shunt insertion.

ELIGIBILITY:
Inclusion Criteria:

* Possible or probable INPH according to the INPH guidelines.
* Symptom duration ≥ 3 months
* Age ≥50 years
* Able to walk 10 meters with or without an assistant device.
* Decision to recommend shunt surgery based either on:

  * Improvement after cerebrospinal fluid (CSF) tap (i.e. positive tap test), or;
  * Increased CSF outflow resistance, or;
  * A combination of "typical" signs/symptoms + "typical" MRI findings;
  * A combination of a-c.

Exclusion Criteria:

* NPH due to hemorrhage, meningitis or stroke (secondary NPH).
* Symptom duration ≥ 5 years.
* Patients considered surgical risk.
* Baseline gait velocity >1.1 m/sec (60 m/min) without assistant device
* Mini Mental State Exam score ≤ 20 points.
* Musculoskeletal condition precluding gait assessment.
* Severe hearing or visual impairment
* Medication in the form of warfarin or novel oral anticoagulant (NOAC)
* Insufficient pressure data below resting pressure during the CSF infusion investigation, i.e. no complete assessment of the pulsatility curve

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in total score on European INPH scale | 3 and 6 months after surgery
  scale describing the cardinal symptoms of INPH
Gait velocity | 3 and 6 months after surgery
  Maximal gait velocity (3 x 10 m)
European INPH scale | baseline (before surgery) and 3 months after surgery
  Change in total score on scale describing the cardinal symptoms of INPH
Gait velocity | baseline (before surgery) and 3 months after surgery
  Maximal gait velocity (3 x 10 m)

SECONDARY OUTCOMES:
Computerized General Neuropsychological INPH Test (CoGNIT) | baseline (before surgery) and 3 months after surgery
  A computerized neuropsychological test battery for use in INPH, which produces a total "neuropsychological" score
Timed up and go test | baseline (before surgery) and 3 months after surgery
  Mobility test: rise from chair, walk 3 m, turn around, walk back and sit down again
EuroQoL's (EQ) standardized 5 dimensions (5D) 5 levels (5L) instrument (EQ-5D-5L™) | baseline (before surgery) and 3 months after surgery
  EuroQoL's standardized instrument for health outcome, which assesses health in 5 dimensions, on 5 levels
Urogenital Distress Inventory (UDI-6) | baseline (before surgery) and 3 months after surgery
  Continence assessment scale
Incontinence Impact Questionnaire, Short Form (IIQ-7) | baseline (before surgery) and 3 months after surgery
  Continence assessment scale
Barthel Index | baseline (before surgery) and 3 months after surgery
  Activities of daily living assessment scale
Modified Rankin scale | baseline (before surgery) and 3 months after surgery
  Disability assessment scale
Geriatric depression scale (GDS-15) | baseline (before surgery) and 3 months after surgery
  Score on a geriatric depression scale consisting of 15 yes/no questions
Mini-mental state examination (MMSE) score | baseline (before surgery) and 3 months after surgery
  Score on the MMSE scale (general mental status)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Malm, MD, PhD, Principal Investigator — Umeå University Hospital; Sara Qvarlander, PhD, Study Director — Umeå University
Locations (5):
- Finland (2):
  - Kuopio university hospital, Kuopio
  - Turku university hospital, Turku
- Sweden (3):
  - Sahlgrenska university hospital, Gothenburg
  - Umeå university hospital, Umeå
  - The Uppsala university hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No